CLINICAL TRIAL: NCT04303754
Title: A Randomized Controlled Trial to Determine the Effects of Diabetes-Specific Formula on Glycemic Control in Individuals With Type 2 Diabetes
Brief Title: Diabetes-Specific Formula in Individuals With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BL45
Record Dates: First submitted 2020-02-22; First posted 2020-03-11 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Bread

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diabetes-Specific Formula (Experimental): Diabetes-Specific Formula
  Interventions: Other: Diabetes-Specific Formula
- Bread and Spread (Experimental): White bread with spread
  Interventions: Other: Bread with Spread
- Rice Porridge (Experimental): Rice Porridge
  Interventions: Other: Rice Porridge

INTERVENTIONS:
Other: Diabetes-Specific Formula — Other: Diabetes Specific Formula
  Arms: Diabetes-Specific Formula
Other: Bread with Spread — Other: White Bread with Spread
  Arms: Bread and Spread
Other: Rice Porridge — Other: Rice Porridge
  Arms: Rice Porridge

SUMMARY:
This study will be conducted using a randomized, controlled, crossover design with three treatments. The purpose of the study is to determine the effects of diabetes-specific formula on glycemic control in individuals with type 2 diabetes.

DETAILED DESCRIPTION:
All study participants will be asked to attend a test session where their glycemic, insulinemic and satiety response to a test meal will be measured, followed by a seven-day washout period where they will not receive or consume any study meal during this period. This cycle will be repeated until all participants complete three test sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 and ≤ 65 years.
2. Participant has type 2 diabetes as evidenced by use of oral antihyperglycemic medication(s), except for DPP-4 inhibitors, with constant dose for at least two months prior to screening and baseline visit. Participant is able to maintain medication number, type and dose throughout the duration of study.
3. Participant with a BMI > 18.5 and ≤ 35.0 kg/m2.
4. Participant is weight stable (has maintained current body weight within 3 kg) for the two months prior to the screening visit.
5. Male or a non-pregnant, non-lactating female, at least 6 weeks postpartum prior to screening visit. A urine pregnancy test is required for all female subjects unless she is not of childbearing potential, defined as postmenopausal for at least one year prior to screening visit or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy). If female is of childbearing potential, is practicing one of the following methods of birth control (and will continue through the duration of the study):

   * Condoms, sponge, diaphragm or intrauterine device;
   * Oral or parenteral contraceptives for 3 months prior to screening visit;
   * Vasectomized partner;
   * Total abstinence from sexual intercourse.
6. If the participant is on a chronic medication such as an anti-hypertensive, lipid-lowering, thyroid medication or hormone therapy, the dosage was constant for at least two months prior to screening and baseline visit. Participant is able to maintain medication number, type and dose throughout the duration of study.
7. Participant is willing to follow protocol as described, including consumption of study product per protocol and completing any forms needed throughout the study.
8. Participant has at least a two-week washout period between completion of a previous research study that required ingestion of any study food or drug and their start in the current study.
9. Participant is willing to refrain from taking non-study diabetes-specific formulas over the entire course of the study.
10. Participant has voluntarily signed and dated an Informed Consent Form (ICF), approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) prior to any participation in the study.

Exclusion Criteria:

1. Participant has a screening HbA1c level <7% or ≥ 10%.
2. Participant uses exogenous insulin or GLP-1 agonists or DPP-4 inhibitors for glucose control.
3. Participant has confirmed type 1 diabetes and/or had history of diabetic ketoacidosis.
4. Participant has current infection (requiring medication), inpatient surgery or received systemic corticosteroid treatment (with the exception of inhaled (includes nasal), topical, and ophthalmic steroids) in the last 3 months; or received antibiotics in the last 3 weeks.
5. Participant has active malignancy (excluding the following dermal malignancies: basal cell carcinoma, squamous cell carcinoma, carcinoma in-situ of the cervix).
6. Participant has significant cardiovascular event within 6 months prior to study entry or history of congestive heart failure.
7. Participant has end stage organ failure (such as end stage renal disease) or was post organ transplant.
8. Participant has a history of renal disease or severe gastroparesis.
9. Participant has current hepatic disease.
10. Participant has had bariatric surgery including gastric balloon; history of gastrointestinal disease (e.g., Crohn's, colitis, celiac) or intestinal surgery that can interfere with consumption or digestion or absorption of study product.
11. Participant has a chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis A, B or C, or HIV.
12. Participant has eating disorder, severe dementia or delirium, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or other conditions that may interfere with study product consumption or compliance with study protocol procedures in the opinion of the principal investigator or study physician.
13. Participant is taking any herbals, dietary supplements, or medications, other than allowed anti-hyperglycemic medications, during the past four weeks prior to screening visit that could profoundly affect (in the opinion of the principal investigator) blood glucose or appetite (examples include orlistat, contrive, qsymia, belviq, incretins, cannabis).
14. Participant uses diabetes-specific formula(s), (e.g. Glucerna, Nestle Nutren Diabetes, Kalbe Diabetasol, Appeton Nutrition Wellness 60+ Diabetic, ForSure, Penta Sure DM, Resurge DM, Diben, Diasip, etc.) defined as more than one eating occasion per week in the last three months.
15. Participant has clotting or bleeding disorders. The use of Plavix® or a similar anticoagulant drug with no reported difficulty during blood draws is allowed and participant is able to maintain medication number, type and dose throughout the duration of study.
16. Participant participates in another study that has not been approved as a concomitant study by AN.
17. Participant has an allergy or intolerance to any ingredient in the study product, as reported by the participant.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose | 4 hours
  Positive area under the curve (AUC) for blood glucose concentration over 0 to 240 minutes.

SECONDARY OUTCOMES:
Postprandial insulin | 4 hours
  Positive area under the curve (AUC) for blood insulin concentration over 0 to 240 minutes.
Appetite | 4 hours
  Appetite (i.e. desire to eat, hunger, prospective consumption, and fullness) will be measured from 0 to 240 minutes using a 100-mm Visual Analogue Scale, anchored with "not at all" on the left side (0 mm) to "extremely" on the right side of the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Siew Ling Tey, Ph.D., Study Chair — Abbott Nutrition; Norlaila Mustafa, MD., Principal Investigator — Universiti Kebangsaan Malaysia Medical Centre
Locations (1):
- Hospital Universiti Kebangsaan Malaysia, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No